CLINICAL TRIAL: NCT01424995
Title: The Natural History of Congenital Trigger Thumbs
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Douglas Hutchinson, M.D., University of Utah
Other Study IDs: 32047
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Congenital Trigger Thumb; Tenosynovitis
Keywords: trigger thumb; flexor pollicis longus tendon of the thumb; stenosis tenosynovitis
MeSH Terms: conditions — Recurrent trigger thumb; Tenosynovitis; Trigger Finger Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This will be a prospective study of all children ages 0 - 5 years old at the time of entry into the study that meet the inclusion criteria who present with congenital trigger thumb. Patient records will be reviewed for eligibility before obtaining parental permission. They will be enrolled in the study at their first visit and followed every year for up to 4 years or until one of the exclusion criteria are met. Participating sites include the University of Utah Orthopaedic Center, Primary Children's Medical Center and Shriners Hospital for Children.

DETAILED DESCRIPTION:
Trigger thumb is a stenosis tenosynovitis of the flexor pollicis longus tendon of the thumb1. The eitiology of congenital trigger thumb is unclear with many authors proposing both hereditary and acquired causes2-4. Surgical release of congenital trigger thumbs has been recommended as definitive treatment, though controversy exists over the natural history of congenital trigger thumbs5-8. There have been a number of studies looking at the natural history of congenital trigger thumbs with spontaneous resolution rates ranging from 0-96% over a median duration of follow up that ranged from 6 months to 48 months9-14. Based on our clinical experience, the investigators do not feel that congenital trigger thumbs resolve spontaneously and that definitive treatment requires surgical release. However, the investigators need to do further scientific research into the natural history of trigger thumbs to determine how often trigger thumb resolves without needing surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital trigger thumb based on physical exam and history, no previous treatment history (either operative or non-operative), no pain associated with the deformity, no functional disability due to the trigger thumb.

Exclusion Criteria:

* Previous operative treatment for the congenital trigger thumb, deformity of the thumb that causes pain, triggering that causes secondary deformity of the thumb, and deformity that prevents normal use of the thumb and hand.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will evaluate all patients who present to our institution with congenital trigger thumb over a one year period and choose not to have a surgical intervention
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2010-12; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The goal of this study is to prospectively evaluate the natural history of congenital trigger thumbs to determine the true incidence of spontaneous resolution. | 4 years
  The following physical exam measurements will be made at the first visit and all subsequent visits until completion of the study: flexion contracture of the interphalangeal joint of both thumbs (resolution of deformity defined as when flexion contracture is 0°), metacarpal-phalangeal joint laxity, and amount interphalangeal joint angular deformity.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas T Hutchinson, MD, Principal Investigator — University of Utah Orthopedics
Locations (1):
- Univeristy of Utah Orthopedic Center, Salt Lake City, Utah, United States